CLINICAL TRIAL: NCT02907489
Title: The Effect of Triple Antibiotic Paste as an Intracanal Medication With an Anti-Inflammatory Drug on Post-Operative Pain of Asymptomatic Uniradicular Necrotic Teeth (A Double Blind Randomized Clinical Trial).
Brief Title: Effect of Triple Antibiotic Paste as an Intracanal Medication With an Anti-Inflammatory Drug on Post-operative Pain.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed omaia ahmed salah, Assistant lecturer in Endodontic departement October 6 University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-194
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Asymptomatic Necrotic Teeth
Keywords: post operative pain; triple antibiotic paste; intracanal medication
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control: Calcium Hydroxide (No Intervention): Non-setting Calcium Hydroxide
- Test: Triple Antibiotic Paste and Anti-Inflammatory Drug (Other): Mixture of ciprofloxacin, metronidazole and minocycline.and diclofenac potassium 50 mg (Catafast)
  Interventions: Other: triple antibiotic paste with an anti-inflammatory drug

INTERVENTIONS:
Other: triple antibiotic paste with an anti-inflammatory drug — Mixture of ciprofloxacin, metronidazole and minocycline.and diclofenac potassium 50 mg (Catafast)
  Arms: Test: Triple Antibiotic Paste and Anti-Inflammatory Drug

SUMMARY:
The purpose of this study is to determine whether the use of triple antibiotic paste as intracanal medication with an anti-inflammatory drug, compared to a calcium hydroxide will reduce postoperative pain and intracanal bacteria or not in patients with asymptomatic necrotic teeth.

DETAILED DESCRIPTION:
This trial is aiming to answer a clinical question whether in patients with asymptomatic necrotic teeth, the use of triple antibiotic paste as intracanal medication with an anti-inflammatory drug, compared to a calcium hydroxide, reduce postoperative pain and intracanal bacteria or not? trial design will be Randomized, controlled, double blinded, unicenter, parallel, two-arm, superiority trial with 1:1 allocation ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age between 18-50 years.
2. Both male and female subjects.
3. Medically free and healthy subjects.
4. Mandibular and maxillary single rooted teeth.
5. Asymptomatic non vital teeth.

Exclusion Criteria:

1. Teeth with acute dentoalveolar abscess.
2. Subjects having more than one tooth that require root canal treatment.
3. Subjects that have taken analgesic, anti-inflammatory or antibiotic drugs during the 10 days prior to the start of treatment.
4. Pregnant females.
5. Subjects with systemic diseases who have endocrine diseases, Infectious diseases or Psychological disturbance.
6. Teeth with periodontal disease or pulp calcification.
7. Subjects taking chronic pain medications.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-10; Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omaia M, Negm M, Nashaat Y, Nabil N, Othman A. The effect of triple antibiotic paste as an intracanal medicament with an anti-inflammatory agent on post-operative pain of asymptomatic uniradicular necrotic teeth: a double blind randomized clinical trial. F1000Res. 2025 Dec 16;8:1687. doi: 10.12688/f1000research.19699.3. eCollection 2019. PMID 41552268
- Available data/document: Study Protocol — https://www.scribd.com/document/328018560/Protocol-Omaia-Repaired-Autosaved

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control: Calcium Hydroxide | Test: Triple Antibiotic Paste and Anti-Inflammatory Drug
Started | 42 | 42
Completed | 40 | 41
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control: Calcium Hydroxide: non setting calcium hydroxide
- Total: Total of all reporting groups
Arm/Group | Control: Calcium Hydroxide | Test: Triple Antibiotic Paste and Anti-Inflammatory Drug | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.23 (9.75) | 32.32 (9.65) | 32.28 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 26 | 20 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain
Description: Visual Analogue Scale (VAS) of post operative pain (The VAS consisted of a 100 mm horizontal ruler without numbers except a "0" at its first part and a "10" in the last part. With "0" indicating the best outcome while "10" the worst outcome. The subjects were asked to mark the point that was equivalent to their pain intensity. The pain levels were classified as no pain [0], mild pain [1-3], moderate pain [4-7] or severe pain [8-10] )
Time Frame: after 24, 48, and 72 hour from the end of the first visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Calcium Hydroxide | Test: Triple Antibiotic Paste and Anti-Inflammatory Drug
Number analyzed (Participants) | 40 | 41
score on a scale
  24 hrs | 3.18 (2.37) | 2.27 (2.28)
  48 hrs | 2.20 (2.00) | 1.39 (1.46)
  72 hrs | 1.30 (1.36) | 0.78 (1.11)
Statistical Analysis 1: Comparison: Control: Calcium Hydroxide vs Test: Triple Antibiotic Paste and Anti-Inflammatory Drug; Test type: Superiority; p = 0.083, Chi-squared — 0.083 for 24 hours, Significant at P ≤ 0.05
Statistical Analysis 2: Comparison: Control: Calcium Hydroxide vs Test: Triple Antibiotic Paste and Anti-Inflammatory Drug; Test type: Superiority; p = 0.041, Chi-squared — 0.041 for 48 hours, Significant at P ≤ 0.05
Statistical Analysis 3: Comparison: Control: Calcium Hydroxide vs Test: Triple Antibiotic Paste and Anti-Inflammatory Drug; Test type: Superiority; p = 0.063, Chi-squared — 0.063 for 72 hours, Significant at P ≤ 0.05

2. Secondary Outcome: Intracanal Bacterial Count
Description: Colony forming units per milliliter of blood agar medium before root canal preparation (S1), after root canal preparation (S2) and after intracanal medication application for 72 hours (S3)
Time Frame: before and after mechanical preparation (at day 0) and after 72 hour from placement of the intracanal medication.
Measure: Mean (Standard Deviation); unit: CFU/ml
Arm/Group | Control: Calcium Hydroxide | Test: Triple Antibiotic Paste and Anti-Inflammatory Drug
Number analyzed (Participants) | 40 | 41
CFU/ml
  S1 | 3.84 (1.70) | 3.85 (2.01)
  S2 | 3.63 (1.63) | 3.36 (1.74)
  S3 | 2.14 (1.36) | 1.33 (1.39)
Statistical Analysis 1: Comparison: Control: Calcium Hydroxide vs Test: Triple Antibiotic Paste and Anti-Inflammatory Drug; Test type: Superiority; p = 0.982, Chi-squared — 0.982 for S1, Significant at P ≤ 0.05
Statistical Analysis 2: Comparison: Control: Calcium Hydroxide vs Test: Triple Antibiotic Paste and Anti-Inflammatory Drug; Test type: Superiority; p = 0.467, Chi-squared — 0.467 for S2, Significant at P ≤ 0.05
Statistical Analysis 3: Comparison: Control: Calcium Hydroxide vs Test: Triple Antibiotic Paste and Anti-Inflammatory Drug; Test type: Superiority; p = 0.01, Chi-squared — 0.01 for S3 Significant at P ≤ 0.05

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control: Calcium Hydroxide | Test: Triple Antibiotic Paste and Anti-Inflammatory Drug
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT02907489/Prot_SAP_000.pdf